CLINICAL TRIAL: NCT00889408
Title: A Phase I Study of DT2219ARL, A Bispecific Singe Chain Immunotoxin for the Treatment of Relapsed or Refractory CD19(+), CD22(+) B-Lineage Leukemia or Lymphoma
Brief Title: DT2219ARL for Relapsed or Refractory CD19 (+), CD 22 (+) B-Lineage Leukemia Or Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012LS075; MT2013-16 (Other: University of Minnesota Blood and Marrow Transplant Program); DT2219ARL
Record Dates: First submitted 2009-04-26; First posted 2009-04-28 (Estimated); Last update posted 2017-12-02 (Actual); Status verified 2017-11

CONDITIONS: Leukemia; Lymphoma
Keywords: refractory chronic lymphocytic leukemia; childhood diffuse large cell lymphoma; childhood grade III lymphomatoid granulomatosis; childhood immunoblastic large cell lymphoma; B-cell adult acute lymphoblastic leukemia; recurrent adult acute lymphoblastic leukemia; B-cell childhood acute lymphoblastic leukemia; recurrent childhood acute lymphoblastic leukemia; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); recurrent adult acute myeloid leukemia; recurrent childhood acute myeloid leukemia; secondary acute myeloid leukemia; B-cell chronic lymphocytic leukemia; relapsing chronic myelogenous leukemia; childhood chronic myelogenous leukemia; cutaneous B-cell non-Hodgkin lymphoma; recurrent adult grade III lymphomatoid granulomatosis; Waldenström macroglobulinemia; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; recurrent childhood grade III lymphomatoid granulomatosis; recurrent childhood large cell lymphoma; recurrent childhood lymphoblastic lymphoma; recurrent childhood small noncleaved cell lymphoma; childhood Burkitt lymphoma; intraocular lymphoma; noncutaneous extranodal lymphoma; prolymphocytic leukemia
MeSH Terms: conditions — Leukemia; Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Large B-Cell, Diffuse; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Congenital Abnormalities; Leukemia, Myeloid, Acute; Waldenstrom Macroglobulinemia; Burkitt Lymphoma; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Dendritic Cell Sarcoma, Interdigitating; Intraocular Lymphoma; Leukemia, Prolymphocytic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): DT2219ARL at assigned dose IV over 4 hours in the outpatient setting on day 1, 3, 5, and 8
  Interventions: Biological: DT2219ARL

INTERVENTIONS:
Biological: DT2219ARL — anti-CD19/CD22 bispecific ligand-directed toxin DT2219ARL

SUMMARY:
This is a phase I dose escalation study of DT2219ARL for the treatment of relapsed or refractory B-lineage leukemia and lymphoma. Patients will receive a single course of DT2219ARL as a 4 hour infusion on days 1, 3, 5, and 8. Weekly follow-up will continue through day 29, at which time a disease reassessment will be done. For patients in remission, follow-up will continue monthly until disease progression or start of a new treatment. Otherwise day 29 will be the final study visit if there is no ongoing toxicity.

This phase I study will use Continual Reassessment Method (CRM) to establish a maximum tolerated dose (MTD) of DT2219ARL. Up to 3 dose levels will be tested with an additional dose level (-1) if dose level 1 proves too toxic. The goal of CRM is to identify the dose level which correspondences to a desired toxicity rate of 33% or less using grade 3 or 4 capillary leak syndrome and any grade 3 or greater toxicity attributed to DT2219ARL as the targeted toxicity (based on CTCAE version 4).

DETAILED DESCRIPTION:
The current study was initially conducted at University of Texas and the Scott and White Cancer Institute (A. Frankel, MD - PI) and M. D. Anderson Cancer Center with 15 evaluable patients enrolled by the end of 2011 (table 1). The 3rd patient enrolled in the 40 μg/kg dose cohort was the first to experience dose limiting toxicity (grade 3 neurological: lower extremity weakness) receiving only 3 of the 4 planned doses. Per study design, the 40 μg/kg would enroll an additional 3 patients to confirm dose limiting toxicity. It is at this point the Texas centers discontinued involvement in the study.

Approximately 15 months after the last patient was enrolled under the original study plan, the protocol was redesigned by the Masonic Cancer Center at the University of Minnesota, building on the experience of the 1st 15 patients enrolled through the Texas centers. To increase efficiency, the study design was changed from the standard 3 x 3 dose escalation to a Continuous Reassessment Method (CRM) model testing 3 doses levels (40, 60, and 80 ug/kg) with an added feature of a dose level -1 (30 ug/kg) in the event dose level 1 proves too toxic. The maximum tolerated dose will be identified once 20 evaluable patients are enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Histologic verification of B-cell lineage leukemia or B cell non-Hodgkin lymphoma and evidence of relapse/refractory disease with the presence of CD19 and/or CD22 by flow cytometry or immunohistochemistry of bone marrow aspirate, peripheral blood or node biopsy
* Disease refractory to conventional therapy and other therapies of higher priority
* Age ≥ 12 years
* Karnofsky Performance status of ≥ 60% or, if less than 16 years of age, Lansky Play Score of ≥ 60 (appendix II)
* Patients must have recovered from effects of prior therapy - at least 2 weeks should have elapsed since the last dose of chemotherapy; however patients who have recovered from the effects of previous treatment and have a >50% rise in peripheral blast count (confirmed twice) or > 50% growth of lymph nodes are immediately eligible - Patients who have relapsed following autologous or allogeneic BMT are eligible
* In order to prevent tumor lysis syndrome, leukemia patients must have a peripheral blast count under 50 x 109/L. This should be achieved with hydroxyurea cytoreduction, prior to starting DT2219ARL as follows - patients with peripheral blasts and a WBC >50 x 109/L, give hydroxyurea 1-5 g daily for up to 5 days to reduce WBC below 50 x 109/L
* Adequate organ function within 14 days (30 days for cardiac and pulmonary) of treatment start defined as:

  * Creatinine: ≤ 1.5 x upper limit of institutional normal (ULN)
  * Hepatic: SGOT (AST) or SGPT (ALT) < 2.5 x ULN and total bilirubin </= 1.5 x ULN
  * General health: Serum albumin ≥ 3.0g/dL
  * Pulmonary: PFTs > 50% if symptomatic or prior known impairment
  * Cardiac: LVEF by ECHO or MUGA ≥ 40%
* Agrees to stay within the Twin Cities metropolitan area (i.e. within 30 miles of the study center) for the duration of the treatment (at least 24 hours after the last dose) and 2) have a capable caregiver
* Women of childbearing potential and men should be advised and agree to practice effective methods of contraception during the course of study
* Voluntary written consent

Exclusion Criteria:

* Presence of leukemic or infectious pulmonary parenchymal disease
* Presence of active CNS leukemia. CSF with <5 WBC/uL will not exclude the patient
* Presence of any uncontrolled systemic infection
* Documented uncontrolled seizure disorder or abnormal neurological examination - a seizure disorder controlled with medication (i.e. no seizures in the previous 6 months) will not exclude a patient
* Documented penicillin or cephalosporin allergies
* Pregnant or lactating - Women of child bearing potential must have a negative pregnancy test within 14 days of study treatment start

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-12-02 (Actual); Primary Completion 2014-07-21 (Actual); Study Completion 2014-07-21 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | 29 days
  This phase I study will use Continual Reassessment method (CRM) method to establish a maximum tolerated dose (MTD) of DT2219ARL when the maximum desired level of toxicity is 33% (defined as grade 3 or 4 capillary leak syndrome toxicities and any grade 3 or greater adverse event attributed to DT2219ARL based on CTCAE v 4).

SECONDARY OUTCOMES:
Therapeutic activity of DT2219ARL | 2 years
  Determined by the change in percentage of blasts in bone marrow and peripheral blood and recovery of normal hematopoiesis and by change in size of lymph nodes/tumor involved by lymphoma

CONTACTS AND LOCATIONS:
Overall Officials: Verokina Bachanova, MD, Principal Investigator — University of Minnesota
Locations (3):
- United States (3):
  - Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas
  - Scott and White Cancer Institute, Temple, Texas